CLINICAL TRIAL: NCT05099653
Title: Study of the Impact of a Physical Activity Programme on the Quality of Life of Patients With Inflammatory Bowel Disease
Acronym: APMICI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Raincy Montfermeil Hospital Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A02807-48
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-10

CONDITIONS: Crohn Disease Haemorrhagic Rectocolitis
Keywords: Physical Activity; Quality of Life
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Comparisons of two parallel groups of patients. The constitution of the two groups will be done by randomisation.
  * A group of 10 to 12 patients with physical activity (protocolised)
  * A group of 10 to 12 patients without physical activity (protocolised)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with physical activity (Experimental): A group of patients with physical activity (protocolized)
  Interventions: Other: physical activity
- patients without physical activity (No Intervention): A group of patients without physical activity (protocolised)

INTERVENTIONS:
Other: physical activity — physical activity
  Arms: patients with physical activity

SUMMARY:
Regular physical activity at a mild to moderate intensity can control inflammation in general and intestinal inflammation in particular during IBD. The effectiveness of a physical activity programme has been evaluated during IBD, but the data are limited to a few studies. Overall, PA improves quality of life but also improves control of disease symptoms and fatigue . The aim of the present work is to evaluate the impact of a physical activity programme on quality of life in patients with IBD. This programme will also evaluate the impact of physical activity on 1) anxiety-depression, 2) fatigue (a frequent and difficult to manage symptom in IBD), 3) IBD activity, 4) smoking cessation.

DETAILED DESCRIPTION:
Crohn's disease and haemorrhagic rectocolitis are Chronic Inflammatory Bowel Diseases (CIBD) which evolve by flare-ups interspersed with periods of remission . The incidence of these two diseases is increasing in France in adults but also and especially in children and adolescents. Indeed, according to data from the EPIMAD registry, from 1988-1990 to 2009-2011, a significant increase in the incidence of both Crohn's disease and haemorrhagic rectocolitis was observed in adolescents (10-16 years): for Crohn's disease from 4.2 to 9.5/10 5 (+126%; P <0.001) and for UC from 1.6 to 4.1/10 5 (+156%; P <0.001). Over the long term, Crohn's disease can progress to intestinal destruction that can be complicated by stricture(s), obstruction(s), fistula(s) and/or abscesses leading to surgical treatment estimated at 50% after 10 years of Crohn's disease progression 1.

Anti-TNFα therapies are widely prescribed for Crohn's disease because they control symptoms, heal the mucosa, reduce hospital admissions and improve quality of life. However, they are associated with side effects often reported by patients, such as asthenia, weight gain and joint pain, symptoms that could be improved by regular physical activity.

Regular physical activity at a mild to moderate intensity can control inflammation in general and intestinal inflammation in particular during IBD. The effectiveness of a physical activity programme has been evaluated during IBD, but the data are limited to a few studies. Overall, PA improves quality of life but also improves control of disease symptoms and fatigue . The aim of the present work is to evaluate the impact of a physical activity programme on quality of life in patients with IBD. This programme will also evaluate the impact of physical activity on 1) anxiety-depression, 2) fatigue (a frequent and difficult to manage symptom in IBD), 3) IBD activity, 4) smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed for IBD in the hospital of Montfermeil
* over 18 years of age
* medical certificate authorising the practice of physical activity
* Informed consent

Exclusion Criteria:

* Age < 18 years
* Medical contraindication to physical activity
* Objection to participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
THE IMPACT OF A PHYSICAL ACTIVITY PROGRAM ON THE QUALITY OF LIFE OF PATIENTS | 6 months
  EVALUATE THE IMPACT OF A PHYSICAL ACTIVITY PROGRAM ON THE QUALITY OF LIFE OF PATIENTS WITH IBD (assessment by IBDQ score)

SECONDARY OUTCOMES:
the impact of the physical activity programme on Psychological state | 6 months
  To measure the impact of the physical activity programme on Psychological state (HAD score)
the impact of the physical activity programme on fatigue (FACIT score) | 6 months
  the impact of the physical activity programme on fatigue (FACIT score)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Nahon, MD, Principal Investigator — Raincy Montfermeil Hospital Group
Locations (1):
- Stéphane Nahon, Montfermeil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Torres J, Mehandru S, Colombel JF, Peyrin-Biroulet L. Crohn's disease. Lancet. 2017 Apr 29;389(10080):1741-1755. doi: 10.1016/S0140-6736(16)31711-1. Epub 2016 Dec 1. PMID 27914655
- [Result] Ungaro R, Mehandru S, Allen PB, Peyrin-Biroulet L, Colombel JF. Ulcerative colitis. Lancet. 2017 Apr 29;389(10080):1756-1770. doi: 10.1016/S0140-6736(16)32126-2. Epub 2016 Dec 1. PMID 27914657
- [Result] Gower-Rousseau C, Vasseur F, Fumery M, Savoye G, Salleron J, Dauchet L, Turck D, Cortot A, Peyrin-Biroulet L, Colombel JF. Epidemiology of inflammatory bowel diseases: new insights from a French population-based registry (EPIMAD). Dig Liver Dis. 2013 Feb;45(2):89-94. doi: 10.1016/j.dld.2012.09.005. Epub 2012 Oct 27. PMID 23107487